CLINICAL TRIAL: NCT00417716
Title: The Efficacy of a Single Intravitreal Injection of Bevacizumab in Patients With Diffuse Diabetic Macular Edema
Brief Title: Use of Intravitreal Bevacizumab in Patients With Diffuse Diabetic Macular Edema
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APEC-0011
Record Dates: First submitted 2006-06-30; First posted 2007-01-04 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus Type 2; Diabetic Macular Edema
Keywords: Diffuse Diabetic Macular Edema; Intravitreal Bevacizumab; Anti-VEGF drugs
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Intravitreal Bevacizumab

SUMMARY:
Intravitreal Bevacizumab is an effective treatment for the diffuse diabetic macular edema

DETAILED DESCRIPTION:
A non-randomized prospective clinical interventional study which includes 45 non previously treated patients with DME. The patients received a single intravitreal injection of 2.5 mg bevacizumab. Follow-up included clinical examination (best corrected visual acuity (BCVA, intraocular pressure (IOP), cataract grading, DME characteristics and systemic check-up) pre-injection, at first visit, at weeks 1 and 2 and months 1 and 3. OCT and fluorescein angiography was evaluated at months 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Macular edema involving the center of the macula demonstrated on OCT
* Clear ocular media
* Untreated patients
* Older than 45 years
* BCVA of the fellow eye at least 20/100

Exclusion Criteria:

* Renal diabetic disease, uncontrolled hypertension or stroke history
* Other ocular disease
* Ocular surgery excepting uncomplicated phacoemulsification
* History of photocoagulation (panretinal or focal)
* History of another intravitreal treatment (like triamcinolone)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09 (Actual); Primary Completion 2005-09 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
BCVA
Fluorescein Angiography
Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Solís-Vivanco, MD, Principal Investigator — Asociación para Evitar la Ceguera en México; Jans Fromow-Guerra, MD PhD, Study Chair — Asociación para Evitar la Ceguera en México; Elizabeth Reyna-Castelán, Study Chair — Asociación para Evitar la Ceguera en México; Juan M Jiménez-Sierra, MD, Study Chair — Asociación para Evitar la Ceguera en México; Myriam Hernández-Rojas, MD, Study Chair — Asociación para Evitar la Ceguera en México; Griselda Alvarez-Rivera, MD, Study Chair — Asociación para Evitar la Ceguera en México; Hugo Quiroz-Mercado, MD, Study Director — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico